CLINICAL TRIAL: NCT01434160
Title: Multi-center, Single-arm Study to Assess the Safety, Efficacy, Discontinuation Rate and Pharmacokinetics of the Low-dose Levonorgestrel Intrauterine Contraceptive System (LCS12) in Post-menarcheal Female Adolescents Under 18 Years of Age for 1 Year, and an Optional 2-year Extension Phase
Brief Title: LCS12 Adolescent Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14371; 2011-002065-37 (EudraCT Number)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Contraception
Keywords: Intrauterine; contraception; adolescent
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Skyla (Levonorgestrel, BAY86-5028)

INTERVENTIONS:
Drug: Skyla (Levonorgestrel, BAY86-5028) — Levonorgestrel intrauterine contraceptive system (LCS12) insertion into the uterus at insertion visit 2 with the study treatment of 12 months. An optional follow up phase up to 3 years will be offered for all subjects completing 12 month treatment time.

SUMMARY:
The study will assess the safety of a sex hormone (levonorgestrel) releasing T-shaped intrauterine contraceptive system in female adolescents under 18 years of age. Approximately 300 generally healthy, post-menarcheal female adolescents with regular menses at the beginning of the study requiring contraception will be enrolled into the study.

Duration of study treatment is approximately 12 months with an option to continue the use of the contraceptive system up to three years if the woman is willing to continue the use after the first 12 months.

The incidence of adverse events over 12 month treatment period will be the main outcome of this study. Also the efficacy (number of pregnancies), discontinuation rate and pharmacokinetics will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed and dated the informed consent form (ICF)
* The subject is female, generally healthy, post-menarcheal, nulliparous or parous, requiring contraception, and is under 18 years of age at the Screening visit
* The subject has regular menstrual cycles without hormonal contraceptive use (at regular intervals of 21-35 days)
* In the opinion of the investigator, the subject has general and uterine conditions suitable for the insertion of levonorgestrel intrauterine contraceptive system (LCS12) (uterine sound depth 6-10 cm)
* Has clinically normal safety laboratory results
* The subject has a normal or clinically insignificant cervical smear (i.e. one that does not require further follow up according to Bethesda or a comparable system)
* The subject is willing and able to attend the scheduled study visits and to comply with the study procedures

Exclusion Criteria:

* Known or suspected pregnancy or is lactating
* Vaginal delivery, cesarean delivery, or abortion less than 6 weeks before Visit 1
* History of ectopic pregnancies
* Infected abortion or postpartum endometritis less than 3 months before Visit 1
* Abnormal uterine bleeding of unknown origin
* Any lower genital tract infection (until successfully treated)
* Acute or history of recurrent pelvic inflammatory disease
* Congenital or acquired uterine anomaly

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse events reported by study subjects | 12 months treatment period
Portion of subjects reporting adverse events | 12 months treatment period

SECONDARY OUTCOMES:
Overall satisfaction rating from 1 to 5 (from very satisfied to very dissatisfied) | 12 months treatment period
Pearl index | 12 months treatment period
Bleeding patterns collected from patients' diary | 12 months treatment period
Concentration of Levonorgestrel in serum | At 1, 3, 6, 9 or 12 months
Concentration of sex hormone binding globulin in serum | At 1, 3, 6, 9 or 12 months
Discontinuation rate | 12 months treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (35):
- Austria (5):
  - Sankt Pölten, Lower Austria
  - Bregenz
  - Vienna
  - Voitsberg
  - Zeltweg
- Belgium (4):
  - Antwerp
  - Bruxelles - Brussel
  - Charleroi
  - Leuven
- Denmark (3):
  - Århus C
  - København NV
  - København S
- Finland (3):
  - Helsinki
  - Kuopio
  - Oulu
- Germany (8):
  - Erlangen, Bavaria
  - Hamburg, Hamburg
  - Cologne, North Rhine-Westphalia
  - Geseke, North Rhine-Westphalia
  - Dippoldiswalde, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Blankenburg, Saxony-Anhalt
- Netherlands (7):
  - Alkmaar
  - Almere Stad
  - Den Helder
  - Enschede
  - Heerlen
  - Nieuwegein
  - Tilburg
- Norway (2):
  - Fornebu
  - Sellebakk
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala

REFERENCES:
- [Derived] Gemzell-Danielsson K, Buhling KJ, Dermout SM, Lukkari-Lax E, Montegriffo E, Apter D. A Phase III, single-arm study of LNG-IUS 8, a low-dose levonorgestrel intrauterine contraceptive system (total content 13.5mg) in postmenarcheal adolescents. Contraception. 2016 Jun;93(6):507-12. doi: 10.1016/j.contraception.2016.02.004. Epub 2016 Feb 9. PMID 26872720